CLINICAL TRIAL: NCT01893983
Title: Motivational Coaching to Enhance Mental Health Engagement in Rural Veterans
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CRE 12-083
Record Dates: First submitted 2013-06-21; First posted 2013-07-09 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-08

CONDITIONS: Mental Health; Rural Health; Veterans Health
Keywords: Mental Health; Veterans Health; Rural; Motivational Interviewing
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Coaching (Experimental): Telephone based Motivational Coaching sessions
  Interventions: Behavioral: Motivational Coaching
- Referral alone (No Intervention): This is the current standard of care

INTERVENTIONS:
Behavioral: Motivational Coaching — Telephone-based Motivational Interviewing aimed at getting Veterans to engage or retain mental health treatment
  Arms: Motivational Coaching

SUMMARY:
The purpose of this study is to investigate health problems among rural Veterans. The research project also aims to test a new telephone-based approach for helping Veterans who need treatment connect with the appropriate care. This study will help us to better understand the kinds of problems Veterans experience. The study will also help us to find better ways to help Veterans get the help they may need.

DETAILED DESCRIPTION:
Project Background: One in five Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF)/Operation New Dawn (OND) Veterans resides in rural areas and primarily receives care from VA Community-Based Outpatient Clinics (CBOCs). Compared to their urban counterparts, rural Veterans experience a significantly greater MH burden and poorer outcomes. Nevertheless, less than 10% of OEF/OIF/OND Veterans with a new PTSD diagnosis attend a minimum number of sessions required for evidence-based treatment, with rurality being one of the strongest predictors of poor engagement. The investigators' pilot study in urban OEF/OIF/OND Veterans demonstrated that telephone Motivational Interviewing (MI) delivered by research staff significantly improved MH treatment initiation and retention in care. However, the investigators do not know whether telephone MI will have as strong an effect on MH treatment engagement when implemented by VA staff in CBOCs serving rural Veterans.

Project Objectives: As a part of the Center for Mental Healthcare and Outcomes Research (CeMOHR) CREATE application to improve rural Veterans' access to evidence-based mental healthcare, the overall goal of this project is to adapt, implement and test an MI-based coaching intervention to improve MH services engagement at CBOCs serving rural Veterans. The specific aims of this project are: (1) Conduct a developmental formative evaluation of perceived barriers to MH treatment engagement and adapt the MI-based treatment engagement intervention and implementation strategy to the needs of stakeholders; (2) Conduct a randomized multi-site pragmatic effectiveness trial comparing MH Referral alone with MH Referral plus MI-based coaching; and (3) Conduct an implementation-focused formative evaluation and use this information to make mid-course corrections to the implementation strategy based on stakeholder and key informant input.

Methods: The investigators will conduct the pragmatic effectiveness trial of the telephone motivational coaching intervention to determine whether, in comparison to MH Referral alone, telephone MI coaching improves MH treatment initiation and retention, the use of e-health MH resources, and perceived need and readiness for and access to MH treatment among rural Veterans who use CBOCs (Aim 2).

Impact: This research will help close the knowledge gap about barriers to care and preferences for MH services among rural Veterans. In addition, information from this project will be used to develop implementation toolkits for MH treatment engagement interventions for rural Veterans. Finally, this project will determine the effectiveness of a telephone Motivational Interviewing engagement intervention using e-health adjuncts, thereby filling a gap in the scientific literature about whether novel interventions can be used by VA staff in CBOCs to overcome rural-urban disparities in MH treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* a Veteran over age 18
* a resident of VISN 16 or 21 catchment areas receiving care at a CBOC with no plans to re-locate within 8 months of enrollment
* positive for 1 or more of the following disorders: PTSD, depression, generalized anxiety disorder, panic disorder, high-risk drinking, and/or illicit substance use

Exclusion Criteria:

* hearing- impaired,
* no working telephone,
* Veterans with self-reported (and/or CPRS-confirmed) diagnoses of schizophrenia, psychosis or bipolar disorder, or active suicidality or homicidality
* received mental health treatment within the last 60 days and/or has future appointments for mental health treatment in the next 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Seal, MD MPH, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koenig CJ, Abraham T, Zamora KA, Hill C, Kelly PA, Uddo M, Hamilton M, Pyne JM, Seal KH. Pre-Implementation Strategies to Adapt and Implement a Veteran Peer Coaching Intervention to Improve Mental Health Treatment Engagement Among Rural Veterans. J Rural Health. 2016 Sep;32(4):418-428. doi: 10.1111/jrh.12201. Epub 2016 Aug 10. PMID 27509291
- [Result] Abraham TH, Koenig CJ, Zamora K, Hill C, Uddo M, Kelly AP, Hamilton MF, Curran GM, Pyne JM, Seal KH. Situating mental health work in place: Qualitative findings from interviews with Veterans in Southeastern Louisiana and Northern California. Health Place. 2017 Sep;47:63-70. doi: 10.1016/j.healthplace.2017.07.001. Epub 2017 Jul 26. PMID 28755653
- See also: Click here for more information about this study: Motivational Coaching to Enhance Mental Health Engagement in Rural Veterans — http://www.vetsreturnhome.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: (1) CBOC providers will refer veterans; (2) VA administrative data will be used to identify veterans; (3) veteran self-referral; (4) "snowball sampling"
Pre-assignment Details: Baseline assessment was used to determine mental health eligibility. Those who did not score high enough on mental health symptoms AND/OR had recently had recently had a mental health visit and/or a schedule mental health visit were excluded.
Period: Overall Study
Arm/Group | Motivational Coaching | Referral Alone
Started | 140 | 140
Completed | 130 | 134
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Population: We baselined 418 participants, 280 were eligible for the study and randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Coaching | Referral Alone | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  years
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 50.1 (13.1) | 51.2 (13.8) | 50.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Female | 27 | 17 | 44
    Male | 112 | 123 | 235
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Hispanic or Latino | 7 | 13 | 20
    Not Hispanic or Latino | 131 | 127 | 258
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    American Indian or Alaska Native | 5 | 3 | 8
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 28 | 36 | 64
    White | 87 | 76 | 163
    More than one race | 8 | 9 | 17
    Unknown or Not Reported | 8 | 15 | 23
Region of Enrollment [Count of Participants; unit: Participants] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  Participants
    United States: number analyzed (Participants) | 139 | 140 | 279
    United States | 139 | 140 | 279
WHOQOL-BREF [Mean (Standard Deviation); unit: units on a scale] — The WHOQOL BREF is a shorter version of the WHO Quality of Life measure that includes four domains: physical health, psychological health, social relationships, and environment domains. The theoretical scale ranges of all 4 domains are the same: 4-20. Higher scores indicate better quality of life. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    Physical Health: number analyzed (Participants) | 139 | 140 | 279
    Physical Health | 12.0 (3.7) | 11.9 (3.3) | 12.0 (3.5)
    Psychological Health: number analyzed (Participants) | 139 | 140 | 279
    Psychological Health | 13.3 (3.1) | 12.9 (2.6) | 13.1 (2.8)
    Social Relationships: number analyzed (Participants) | 139 | 140 | 279
    Social Relationships | 13.0 (4.2) | 12.7 (4.0) | 12.8 (4.1)
    Environment: number analyzed (Participants) | 139 | 140 | 279
    Environment | 14.6 (2.9) | 14.1 (2.9) | 14.3 (2.9)
Mental Health Treatment Experiences in the last 5 years [Count of Participants; unit: Participants] — Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  Participants
    Primary Care: number analyzed (Participants) | 139 | 140 | 279
    Primary Care | 50 | 43 | 93
    Mental Health- Individual or Group Counseling: number analyzed (Participants) | 139 | 140 | 279
    Mental Health- Individual or Group Counseling | 73 | 76 | 149
    Substance Abuse Treatment: number analyzed (Participants) | 139 | 140 | 279
    Substance Abuse Treatment | 8 | 12 | 20
    Inpatient Psychiatric Treatment: number analyzed (Participants) | 139 | 140 | 279
    Inpatient Psychiatric Treatment | 5 | 5 | 10
    Counseling by Social Worker: number analyzed (Participants) | 139 | 140 | 279
    Counseling by Social Worker | 19 | 18 | 37
    Counseling by chaplain or other religious person: number analyzed (Participants) | 139 | 140 | 279
    Counseling by chaplain or other religious person | 6 | 10 | 16
    Marital, relationship or family counseling: number analyzed (Participants) | 139 | 140 | 279
    Marital, relationship or family counseling | 13 | 8 | 21
    Self-help group: number analyzed (Participants) | 139 | 140 | 279
    Self-help group | 10 | 5 | 15
    Internet/Mobile Application treatment program/supp: number analyzed (Participants) | 139 | 140 | 279
    Internet/Mobile Application treatment program/supp | 9 | 10 | 19
    Telephone counseling program: number analyzed (Participants) | 139 | 140 | 279
    Telephone counseling program | 10 | 16 | 26
    Psychiatric medication: number analyzed (Participants) | 139 | 140 | 279
    Psychiatric medication | 81 | 85 | 166
    Research study: number analyzed (Participants) | 139 | 140 | 279
    Research study | 7 | 4 | 11
Readiness Ruler: Assessment of Motivation for Treatment [Mean (Standard Deviation); unit: units on a scale] — All 3 measures have a range of 0-10 for both arms.
  The higher scores are the better. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    How important is it for you to receive treatment r: number analyzed (Participants) | 139 | 140 | 279
    How important is it for you to receive treatment r | 5.2 (3.1) | 5.9 (3.5) | 5.5 (3.3)
    How confident are you that you would get treatment | 5.9 (3.4) | 6.4 (3.3) | 6.1 (3.4)
    How ready are you to receive treatment right now f | 6.2 (3.3) | 6.9 (3.4) | 6.6 (3.4)
Severity Measure for Depression-Adult (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The theoretical scale range is 0-27, with higher scores indicating greater severity of depression. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 11.3 (6.1) | 12.2 (5.9) | 11.8 (6.0)
Severity Measure for Generalized Anxiety Disorder-Adult [Mean (Standard Deviation); unit: units on a scale] — The investigators used the averaged total score calculated by dividing the raw total score by number of items in the measure. The theoretical scale range is 0-4, with higher scores indicating greater severity of anxiety disorder. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 1.5 (0.9) | 1.5 (0.9) | 1.5 (0.9)
Severity Measure for Panic Disorder-Adult [Mean (Standard Deviation); unit: units on a scale] — The investigators used the averaged total score calculated by dividing the raw total score by number of items in the measure. The theoretical scale range is 0-4, with higher scores indicating greater severity of panic disorder. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 0.8 (1.0) | 0.9 (1.0) | 0.8 (1.0)
PCL-5 [Mean (Standard Deviation); unit: units on a scale] — PCL-5 is the PTSD Checklist for DSM-5. It is a 20-item self-report measure that assesses 20 symptoms of PTSD. Each item is on a 5-point Likert scale ranging from 0-4, and the total score range is 0-80, with the higher scores indicating more severe PTSD symptoms. A cut-point score of 33 is considered as a diagnostic criterion for PTSD.
  In our study, we did not intend to diagnose PTSD. Instead, we simply compared total scores of PCL-5 between two arms. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 25.0 (19.0) | 27.6 (18.1) | 26.3 (18.6)
WHO - ASSIST V3 [Mean (Standard Deviation); unit: units on a scale] — Ranges of scores:
  tobacco: 0-31, alcohol: 0-39, cannabis: 0-39, cocaine: 0-39, amphetamine: 0-39, inhalants: 0-39, sedatives: 0-39, hallucinogens: 0-39, opioid: 0-39.
  The higher scores indicate worse outcome. Population: One participant from the motivational coaching arm withdrew and requested their data not be used in data analysis.
  units on a scale
    Tobacco: number analyzed (Participants) | 139 | 140 | 279
    Tobacco | 8.6 (9.9) | 8.3 (9.9) | 8.5 (9.9)
    Alcohol: number analyzed (Participants) | 139 | 140 | 279
    Alcohol | 7.8 (8.4) | 7.6 (8.7) | 7.7 (8.5)
    Cannabis: number analyzed (Participants) | 139 | 140 | 279
    Cannabis | 3.2 (4.8) | 3.5 (6.0) | 3.3 (5.4)
    Cocaine: number analyzed (Participants) | 139 | 140 | 279
    Cocaine | 0.5 (2.5) | 0.8 (3.3) | 0.7 (2.9)
    Amphetamine: number analyzed (Participants) | 139 | 140 | 279
    Amphetamine | 0.2 (0.9) | 0.5 (1.6) | 0.4 (1.3)
    Inhalants: number analyzed (Participants) | 139 | 140 | 279
    Inhalants | 0.01 (0.2) | 0.2 (1.6) | 0.1 (1.1)
    Sedatives: number analyzed (Participants) | 139 | 140 | 279
    Sedatives | 0.8 (4.1) | 0.4 (2.1) | 0.6 (3.3)
    Hallucinogens: number analyzed (Participants) | 139 | 140 | 279
    Hallucinogens | 0.1 (0.4) | 0.2 (0.6) | 0.1 (0.5)
    Opioids: number analyzed (Participants) | 139 | 140 | 279
    Opioids | 0.2 (2.5) | 0.9 (4.0) | 0.6 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Mental Health (MH) Treatment Engagement
Description: Motivational Coaching (vs. Control) on MH treatment initiation. This will be measured by self-report and by checking the subjects medical record. The investigators will adjust by clustering for CBOC and region as well as potential confounding by other covariates
Time Frame: 26 months
Population: Including 272 patients who provided primary outcome data (excluding those who withdrew).
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Coaching | Referral Alone
Number analyzed (Participants) | 137 | 135
Participants | 78 | 74
Statistical Analysis 1: Comparison: Motivational Coaching vs Referral Alone; Compare 2 groups in regard to time to first mental health treatment using Cox proportional hazards regression; Test type: Equivalence — Compare whether 2 groups had any difference in risk/hazard of mental health engagement at any time during follow-up; p = 0.660, Regression, Cox — P value 0.05 is the threshold for statistical significance; Adjusted for site, mental health treatment history and mental health symptom severity at baseline, baseline amphetamine and opioid scores; Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.81 to 1.58] — The referral alone arm is the reference group (denominator), and the motivational coaching arm is the numerator

2. Secondary Outcome: Mental Health (MH) Treatment Retention
Description: Motivational Coaching (vs. Control) on MH treatment retention. This will be measured by self-report and by checking the subjects medical record. The investigators will adjust by clustering for CBOC and region as well as potential confounding by other covariates
Time Frame: 26 months
Population: Including patients who provided primary outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Coaching | Referral Alone
Number analyzed (Participants) | 137 | 135
Participants | 67 | 62

3. Other Pre Specified Outcome: Mental Health Symptoms, Substance Use Scores and Quality of Life (QOL) Measures.
Description: Depression, anxiety, panic, PTSD, tobacco, alcohol, cannabis, cocaine, amphetamine, inhalants, sedatives, hallucinogen, opioid, and QOL domains: physical health, psychological health, social relationships, and environment.
  Ranges of scores: depression: 0-27, anxiety: 0-4, panic: 0-4, PTSD: PTSD: 0-80., tobacco: 0-31, alcohol: 0-39, cannabis use: 0-39, cocaine: 0-39, amphetamine: 0-39, inhalants: 0-39, sedatives: 0-39, hallucinogen: 0-39, opioid: 0-39, QOL physical health: 4-20, QOL psychological health: 4-20, QOL social relationships: 4-20, QOL environment: 4-20.
  Higher scores mean worse outcomes for mental health symptoms and substance use scores; higher scores mean worse outcomes for quality of life measures.
Time Frame: 26 months
Population: Including patients who reported mental health symptoms, substance use, and quality of life.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Coaching | Referral Alone
Number analyzed (Participants) | 102 | 118
score on a scale
  depression | 9.4 (6.2) | 11.1 (6.5)
  anxiety | 1.2 (0.9) | 1.3 (0.8)
  panic | 0.6 (0.9) | 0.7 (0.9)
  PTSD | 25.1 (18.4) | 29.7 (16.7)
  tobacco | 8.8 (9.5) | 9.2 (10.0)
  alcohol | 7.1 (7.7) | 7.7 (8.6)
  cannabis | 3.1 (4.8) | 4.6 (6.7)
  cocaine | 0.7 (2.9) | 0.9 (2.5)
  amphetamine | 0.3 (1.6) | 0.7 (2.5)
  inhalants | 0 (0) | 0.2 (1.4)
  sedatives | 0.5 (2.9) | 0.8 (3.1)
  halluninogens | 0.2 (1.1) | 0.2 (0.8)
  opioid | 0.5 (2.7) | 0.9 (3.8)
  QOL physical health domain | 12.6 (3.7) | 12.0 (3.1)
  QOL psychological health domain | 13.4 (2.8) | 12.7 (2.5)
  QOL social relationships domain | 13.3 (3.9) | 12.1 (3.8)
  QOL environment domain | 14.4 (2.5) | 13.6 (2.6)

4. Other Pre Specified Outcome: Self-care Activities
Description: Five types of self-care activities to relieve stress: internet or mobile applications, community groups (church groups, gun clubs), community classes (Yoga, cooking), alternative treatments (acupuncture, chiropractor, massage), and other self-care activities (meditation, fishing, walking).
Time Frame: 26 months
Population: Including participants who responded to survey questions during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Coaching | Referral Alone
Number analyzed (Participants) | 115 | 120
Participants
  Internet or mobile applications | 84 | 63
  Community groups | 59 | 52
  Community classes | 31 | 16
  Alternative treatments | 40 | 38
  Self-care activities | 111 | 109

ADVERSE EVENTS:
Time Frame: 2 years and 9 months
Description: Adverse events were collected during telephone interactions only if reported by the participant.
Arm/Group | Motivational Coaching | Referral Alone
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/140
Serious Adverse Events (participants affected / at risk) | 3/140 | 2/140
Other Adverse Events (participants affected / at risk) | 4/140 | 2/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Coaching (N=140) | Referral Alone (N=140)
Hospitalization from Car Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — He was involved in a car accident and hospitalized, suffering a broken arm and a facial injury. He said he was too upset with the VA to continue in the study.
Hospitalization from Stomach Flu (Gastrointestinal disorders) | 0 (0) | 1 (1) — She's been having a stomach illness, was totally out of it and had to go to urgent care/hospital get to get fluids etc. It sounded like a pure stomach virus, with all the sxs.
Hospitalization for Lung Transplant (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — The veteran was in the hospital for a lung transplant. She self reported that she has been in the hospital for about 3 weeks. At a future interview she was hospitalized again due to complication related to the lung transplant.
Hospitalization for Abdominal Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Participant had abdominal surgery
Hospitalization due to injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant stated that he had been assaulted/beaten by another veteran. This assault required a 4-day hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Coaching (N=140) | Referral Alone (N=140)
Lung Cancer Diagnosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant stated that he had been diagnosed with lung cancer a few months prior
Hurt Shoulder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant stated that he hurt his should in previous week and had to have an MRI
Recently illness (Infections and infestations) | 1 (1) | 0 (0) — Participant self reported that he has been ill the last three weeks. He did not see the doctor for this event, and says it is starting to break away from him now. He said he was not sure if it was cold or flu, but is not running a fever.
Adverse Events related to PTSD (Psychiatric disorders) | 1 (1) | 0 (0) — Participant claims that since they have been talking about their MH issues and prior trauma, the participant's drinking and gambling has increased, and they are experiencing more dreams about her trauma.
Broken Rib (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant stated that he had broken a rib while at work
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — Participant called PI to explain that he was very concerned about the personal information that he provided in this study and the security of that data. These concerns have caused him lots of anxiety and he has lost sleep over this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT01893983/Prot_SAP_000.pdf